CLINICAL TRIAL: NCT04841200
Title: Effects of Chinese Medicine on Patients With Coal Worker's Pneumoconiosis: Study Protocol for a Randomized Controlled Trial
Brief Title: TCM for Coal Worker's Pneumoconiosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TCM for CWP
Record Dates: First submitted 2021-04-05; First posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2020-12

CONDITIONS: Coal Worker's Pneumoconiosis
Keywords: Coal Worker's Pneumoconiosis; RCT; TCM
MeSH Terms: conditions — Anthracosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chinese medicine compound combined with symptomatic treatments (Experimental): Patients in this arm will receive Chinese medicine compound based on TCM syndrome differentiation in addition to symptomatic treatments.
  Interventions: Drug: Chinese medicine compound combined with symptomatic treatments
- Chinese medicine compound placebod combined with symptomatic treatments (Placebo Comparator): Patients in this arm will receive Chinese medicine compound placebo based on TCM syndrome differentiation in addition to symptomatic treatments.
  Interventions: Drug: Chinese medicine compound placebo combined with symptomatic treatments

INTERVENTIONS:
Drug: Chinese medicine compound combined with symptomatic treatments — All patients were given symptomatic treatment according to consensus of Chinese experts on pneumoconiosis treatment (2018).
  There are 3 Recipe for the 3 traditional Chinese syndrome.
  Yang Qing Chen Fei Granules for syndrome of yin deficiency and heat-dryness, Bao Jin Chen Fei Granules for syndrome of pulmonary qi deficiency, Jin Shui Chen Fei Granules syndrome of deficiency of pulmonary and renal qi
  All drugs were made into granules by Sichuan Neo-Green Pharmaceutical Technology Development Co., Ltd.
  Each type of granule will be given orally, twice a day, for 52 weeks.
  Arms: Chinese medicine compound combined with symptomatic treatments
Drug: Chinese medicine compound placebo combined with symptomatic treatments — All patients were given symptomatic treatment according to consensus of Chinese experts on pneumoconiosis treatment (2018).
  There are 3 placebo Recipe for the 3 traditional Chinese syndrome.
  Yang Qing Chen Fei Granules placebo for syndrome of yin deficiency and heat-dryness, Bao Jin Chen Fei Granules placebo for syndrome of pulmonary qi deficiency, Jin Shui Chen Fei Granules placebo for syndrome of deficiency of pulmonary and renal qi
  All drugs were made into granules by Sichuan Neo-Green Pharmaceutical Technology Development Co., Ltd. The appearance, shape, color and packaging of Chinese medicine compound placebo are the same as those of drugs.
  Each type of granule will be given orally, twice a day, for 52 weeks.
  Arms: Chinese medicine compound placebod combined with symptomatic treatments

SUMMARY:
This study aims to evaluate the clinical efficacy of traditional Chinese medicine in the treatment of pneumoconiosis and to provide high-quality evidence for the prevention and treatment of pneumoconiosis.

DETAILED DESCRIPTION:
Pneumoconiosis refers to a group of occupational lung diseases characterized by diffuse fibrosis of the lung tissue. It is caused mainly by long-term inhalation and deposition of mineral dust, with varying levels of pathogenicity, into the lungs during occupational activities. Currently, there are a lack of effective therpy options for pneumoconiosis. Traditional Chinese Medicine (TCM) present a favorable prospect in treating pneumoconiosis. But the quality of the research was low. This needs to be further investigated by well-designed RCT to demonstrate the effect of TCM for pneumoconiosis.

In this study, a multicenter, randomized, double-blind, parallel controlled trial was designed. Patients with coal worker's pneumoconiosis were randomly divided into treatment group and control group by central random distribution system. For the treatment group, which was given symptomatic treatments, patients were additionally given Chinese medicine compound based on TCM syndrome differentiation. For the control group, which was given symptomatic treatments, patients were additionally given Chinese medicine compound placebo based on TCM syndrome differentiation. The intervention course is 52 weeks.The Six-minute Walking Distance (6MWD) and the Chronic Obstructive Pulmonary Disease Assessment Test (CAT) score were taken as the primary outcomes, while the Modified British Medical Research Council Dyspnea Scale (mMRC) score, Pulmonary function, Clinical symptoms and signs questionnaire, the Hospital Anxiety and Depression Scale (HADS) score, and the Short Form 36 Health Survey Questionnaire (SF-36) score as the secondary outcomes, third-party data management and blind evaluation were adopted.

ELIGIBILITY:
Inclusion Criteria:

1. Pneumoconiosis (coal workers' pneumoconiosis) patients aged 18 to 75 years;
2. Comply with TCM syndrome differentiation standards;
3. Sign informed consent forms.

Exclusion Criteria:

1. Patients who do not get rid of the dust;
2. Patients with active tuberculosis, idiopathic pulmonary fibrosis, asthma, bronchiectasis, pulmonary embolism, chronic respiratory failure or other severe respiratory diseases;
3. Acute exacerbations occurred within 1 month before selection;
4. Patients with severe cardiovascular and cerebrovascular diseases (malignant arrhythmia, unstable angina, acute myocardial infarction, HF New York Heart Association classes III to IV, stroke, cerebral hemorrhage);
5. Patients with severe liver and kidney disease (liver cirrhosis, portal hypertension, dialysis, kidney transplantation);
6. Tumor patients undergoing resection, radiotherapy and chemotherapy within 5 years before selection;
7. Patients with activity difficulties caused by neuromuscular diseases;
8. Patients with severe arthritis;
9. Patients with severe peripheral vascular disease;
10. Pregnant and lactating women;
11. Patients with severe cognitive and mental disorders;
12. Clinical investigators who are participating in other interventions within 1 month before selection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2021-04-15 (Estimated); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
COPD assessment test (CAT) | Change from baseline CAT scores at week 13, 26, 39, and 52.
  The COPD assessment test (CAT) is a self-administered questionnaire that measures health-related quality of life. It is an 8-item questionnaire on a 0-5 point scale with higher values indicating greater impact of COPD. The item response values of CAT are summed to produce a single score that ranges from 0-9 (low impact), 10-20 (medium impact), 21-30 (high impact) and 31-40 (very high impact).
Six-minute walk distance (6MWD) | Change from baseline 6MWD at week 13, 26, 39, and 52.
  Six-minute walk distance (6MWD) will be conducted to assess exercise capacity.

SECONDARY OUTCOMES:
modified Medical Research Council (mMRC) | Change from baseline mMRC scores at week 13, 26, 39, and 52.
  The modified Medical Research Council (mMRC) scale is a 5-point (0-4) scale based on the severity of dyspnoea. "0" means no dyspnea perception, "4" means severe dyspnea perception.
Pulmonary Function | Changes from baseline to week 26, and 52 in pulmonary function parameters [FEV1 (L),FVC (L),FEV1/FVC (%),FEV1%,PEF (L/sec),DLCO (mL/mmHg/min)]
  Pulmonary functions were measured with spirometric tests by experienced physical therapists.
Clinical Symptoms and Signs Questionnaire | Change from baseline clinical symptoms and signs questionnaire scores at week 13, 26, 39, and 52.
  Assessment will be performed by clinical symptoms and signs questionnaire. The clinical symptoms to be evaluated in this study include cough, expectoration, chest tightness, shortness of breath, wheezing and cyanosis. A score of 0-3 will be given to every symptom or sign with a higher score indicating a worse conditoin.
MOS 36-Item Short-Form Health Survey (SF-36) | Change from baseline SF-36 scores at week 13, 26, 39, and 52.
  The MOS 36-Item Short-Form Health Survey (SF-36) is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 items, divided into eight areas: functional capacity, physical aspects, pain, health general state, vitality, social aspects, emotional aspects, mental health and one question of comparative evaluation between current health conditions and the health conditions from the previous year. Scores range from 0 to 100 where zero corresponds to the "the worst health state" and 100, to "the best health state".
Hospital Anxiety and Depression Scale (HADS) | Change from baseline HADS scores at week 13, 26, 39, and 52.
  Hospital Anxiety and Depression Scale (HADS) questionnaire. The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The anxiety and depression subscales each range from 0 to 21, with higher scores indicating higher anxiety/depression complains. Patients were defined as having anxiety or depression or both if the score was 8 or more in the corresponding subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-sheng Li, Professor, Study Chair — The First Affiliated Hospital of Henan University of Traditional Chinese Medicine
Locations (1):
- The First Affiliated Hospital of Henan University of Traditional Chinese Medicine, Zhengzhou, Henan, China